CLINICAL TRIAL: NCT04524494
Title: Human Intestinal Amino Acid Absorption and the Role of a Local (Renin)-Angiotensin System (RAS)
Brief Title: Human Intestinal Amino Acid Absorption and the Role of a Local RAS
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: EK1744; ks20Vuille
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Renin-Angiotensin Aldosterone System (RAS)
Keywords: Renin Angiotensin System; Angiotensin Converting Enzyme 2 (ACE2); Angiotensin II AT1 Receptor Blocker; ACE inhibitors; intestinal amino acid absorption
MeSH Terms: interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — intestinal tissue samples blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAS- active medication: Patients taking RAS- active medication (ACE- Inhibitor, Angiotensin II AT1 Antagonist (Sartan)) on a daily Basis for at least 6 months for medical reasons
  Interventions: Other: biopsy of intestinal tissue; Other: blood draw; Other: urine collection
- no RAS- active medication: Patients not taking RAS- active medication
  Interventions: Other: biopsy of intestinal tissue; Other: blood draw; Other: urine collection

INTERVENTIONS:
Other: biopsy of intestinal tissue — 4 intestinal tissue biopsies taken from descending Duodenum, 2 intestinal tissue biopsies taken from Ileum, 2 intestinal tissue biopsies taken from ascending colon (additional to routine biopsies taken for gastrointestinal diagnostic)
Other: blood draw — 40 ml blood draw (in Heparin blood tubes) (additional to routine blood draw taken for gastrointestinal diagnostic)
Other: urine collection — Midstream Urine collection

SUMMARY:
This study is to find out what role a local intestinal RAS (renin angiotensin system) plays in the context of amino acid absorption in the human intestinal tract and how this RAS and thus the amino acid absorption is influenced by the RAS-active drugs (angiotensin II AT1 receptor blockers (sartans) or ACE inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 18-35 kg/m2
* cohort 1: therapy with an angiotensin II AT1 antagonist or ACE Inhibitor
* cohort 2: no therapy with an angiotensin II AT1 antagonist or ACE Inhibitor
* Carrying out a diagnostic gastroscopy, colonoscopy or a combined gastroscopy / colonoscopy
* Existence of written consent after detailed information about the study

Exclusion Criteria:

* Severe pathological changes in the gastrointestinal tract (e.g. sprue, stomach ulcers, malignancies); (reflux esophagitis and gastritis are not Exclusion criteria)
* History of gastrointestinal tract surgery (except for appendectomy and inguinal hernia surgery)
* History of malignancy
* Severe acute and chronic organ diseases requiring treatment (e.g. kidney replacement therapy)
* Patients with an increased risk of bleeding (e.g. oral anticoagulation, coagulation disorders)
* Drug or alcohol abuse
* Mental impairment limiting the ability to meet all study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undertaking a gastroscopy and / or colonoscopy for a medical indication
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01-27 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-05-31 (Actual)

PRIMARY OUTCOMES:
messenger ribonucleic acid (mRNA) quantification in intestinal tissue biopsy | single time-point at baseline
  mRNA quantification in intestinal tissue biopsy: mRNA content coding for regulatory RAS protein is measured relative to the mRNA content, which codes for the structural protein villin.
amino acid concentration in blood sample | single time-point at baseline
  amino acid concentration in blood sample by High Performance Liquid Chromatography (HPLC)
amino acid concentration in urine sample | single time-point at baseline
  amino acid concentration in urine sample by HPLC (High Performance Liquid Chromatography)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael N Vuille-dit-Bille, Dr. med., Principal Investigator — Universitäts-Kinderspital beider Basel (UKBB)
Locations (2):
- Switzerland (2):
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - UniversitätsSpital Zürich, Zurich